CLINICAL TRIAL: NCT06559293
Title: Pilot Feasibility Study of Laryngeal Ultrasound in the Paediatric Population
Brief Title: Pilot Feasibility Study of Laryngeal Ultrasound in the Paediatric Population - ECHO LARYNX
Acronym: ECHO-LARYNX
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/86
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Laryngeal Diseases; Ultrasound
Keywords: transcutaneous laryngeal ultrasound; pediatric population; otorhinolaryngology; ENT
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laryngeal ultrasound — laryngeal ultrasound with linear probe will be positioned on the patient's neck. A list of anatomical sites to be visualised will be determined beforehand. Once all the pre-determined structures have been visualised, in an axial and sagittal plane, we will note the position of the ultrasound probe and its orientation. This will enable us to determine the ideal position of the ultrasound probe for obtaining all the elements of interest on a section that will be called the reference section.

SUMMARY:
Nasofibroscopy is the gold standard for laryngeal pathology diagnosis. However, this examination is invasive and can be poorly tolerated in the pediatric population. Laryngeal ultrasound appears to be a better tolerated alternative. However, few data exist in the pediatric population in the literature. The aim of this study is to evaluate the feasibility of laryngeal ultrasound in a larger pediatric population of pathological and non-pathological subjects.

DETAILED DESCRIPTION:
According to current knowledge, the gold standard for diagnosing laryngeal pathologies is flexible fiberoptic laryngoscopy (FFL), as it allows visualisation of the motricity of the laryngeal structures and the appearance of the mucous membranes. However, this is an invasive examination, which can be poorly tolerated in the pediatric population. This poor tolerance can make it difficult to obtain an accurate diagnosis because of the child's movements. With the aim of improving patient comfort without compromising diagnostic performance, some studies describe laryngeal ultrasound (LUS) as an alternative to FFL. This imaging examination appears to be better tolerated than FFL because it is less invasive for the patient. However, there are few data available in the infant population. The main limitations of LUS are obtaining a satisfactory ultrasound window and inter-rater reproducibility. For these reasons, the aim of this study is to assess the feasibility of LUS in the pediatric population and to obtain reference frame enabling the different laryngeal structures to be visualised. We will include around one hundred patients treated in the pediatric ENT unit, with or without laryngeal pathology. An ultrasound record will be performed during the consultation in addition to the usual examination. The record will be analysed by a blinded assessor. A single consultation will be required and no follow-up is planned.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in the pediatric ENT unit at Bordeaux University Hospital, aged between 0 and 15 years

Exclusion Criteria:

* intubated patient,
* haemodynamic
* respiratory instability
* opposition to participation expressed by parents or patient

Ages: 0 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Patients treated in the pediatric ENT department at Bordeaux University Hospital, whether in consultation hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Reproducible ultrasound images | At Baseline (D0)
  Define detailed and reproducible ultrasound images using consistent anatomical landmarks for diagnostic assessment of the larynx

SECONDARY OUTCOMES:
Demographic characteristics | At Baseline (D0)
  We will evaluate the demographic characteristics that may affect the reproducibility of ultrasound images

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SAGARDOY, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Hôpital Pellegrin, Service d'oto-rhino-laryngologie, de chirurgie cervico-faciale et d'ORL pédiatrique, Bordeaux, France